CLINICAL TRIAL: NCT06548386
Title: Feasibility and Accuracy of a Novel Pleural Drain Gas Analyzer in Detecting Air Leaks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lung Healing Technologies Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000003
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Air Leak From Lung; Pneumothorax
Keywords: alveolopleural fistula
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Pleural gas analysis — Patients enrolled in this study will undergo both VI and pleural gas analysis to assess for air leak following surgical chest tube placement.
  For pleural gas analysis, an outlet gas analyzer will be kept on the outlet port of the chest drain for the entire duration of time that a chest tube is in place. We plan to collect both continuous data, looking for intermittent spikes and gas changes, along with episodic data collected during specific air leak assessments. The gas analyzer may better be able to measure an air leak during these specific procedures conducted twice per day, but it will also be used at the outlet port of the chest drain the rest of the time to continuously check for an air leak throughout the hospital stay.

SUMMARY:
The goal of this study is to assess the clinical feasibility of a novel, reusable, low cost gas analyzer that detects breath in chest drains in order to diagnose and heal air leaks. The investigators have developed prototype gas analyzers that attach to the outlet of any analog chest drain, and can be connected temporarily to the sampling port. They detect breath by measuring CO2, O2, and pressure, in order to supplement the information provided by the bubbles in the water seal.

DETAILED DESCRIPTION:
Tests on patients in 2013 at Northwestern demonstrated that gas analysis can help diagnose and heal air leaks by detecting breath in chest drains, as documented in the investigator's patents and peer-reviewed publications. CO2 is 100 times higher in the lung than ambient, and O2 the same amount lower in ppm. The length of time that it takes to detect breath at the outlet is related to the size of the air leak. O2 is available next to every bed, often used in recovery, and when high O2 is quickly detected at the sampling port, the only source can be an active air leak.

The primary aim is to assess whether the device can accurately measure changes in gas flow from an analog pleural drain and whether this accurately detects pleural air leaks.

Specific aim 1: To determine whether the gas analyzer device can measure changes in exhaled gas levels and if this can distinguish true air leaks from false air leaks.

Sub aim 1: Assess how patient characteristics such as extent of resection, pre-existing conditions such as COD, lung function test, etc, affect the efficacy of the device.

Specific aim 2: Compare the accuracy of pleural air leak measured via gas analysis to the accuracy of pleural air leak detection as measured by standard VI.

The hypothesis is that the prototype pleural gas analyzer, through detection of carbon dioxide and oxygen levels, can distinguish true air leaks from false air leaks more accurately than the traditionally practiced method of Visual Inspection of bubbles in the chest drainage unit (VI).

Study Endpoints:

The primary end point of this study is detection of air leak, either by VI or prototype pleural gas analysis.

True Air Leak Definition:

1. Both visual inspection and pleural gas analysis demonstrate an air leak
2. Development of a pneumothorax at any point up to 4 weeks after chest tube removal
3. Pneumothorax develops during a clamp trial to assess for true air leak (failed clamp trial)
4. Patient discharged home with chest tube due to clinical concern (even in absence of clamp trial) of ongoing air leak
5. Development of clinically significant subcutaneous emphysema either with a chest tube in place or after chest tube removal (defined as an increase beyond initial post op, observable to patient or care team) Secondary endpoint is comparison in accuracy in detection of air leak between VI and gas analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled for thoracic surgery and expected to have chest tube placed
2. For patients who are unable to sign consent, but meet all of the inclusion criteria and none of the exclusion criteria, a legally appointed representative (LAR) will be allowed to sign consent for that patient
3. Patients that provide informed consent for the study
4. Patients >18 years old

Exclusion Criteria:

1. Patients with hemodynamic instability
2. Pregnant patients
3. Prisoners
4. Individuals who are not yet adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy alone | One year
  Whether gas analysis can accurately assess for air leak

SECONDARY OUTCOMES:
Using VI as well | One year
  Comparison of accuracy in air leak assessment between gas analysis and visual inspection

CONTACTS AND LOCATIONS:
Locations (1):
- Endeavor Health, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No